CLINICAL TRIAL: NCT06185660
Title: A National, Multicenter, Prospective, Observational Study to Assess Patient Characteristics, Treatment Algorithms and Disease Management of Hyperkalaemia Patients With Chronic Kidney Disease or Under Dialysis or With Heart Failure, Treated With Sodium Zirconium Cyclosilicate in Greece
Acronym: SHIELD
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9480R00055
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Hyperkalaemia
Keywords: Hyperkalaemia
MeSH Terms: conditions — Hyperkalemia | interventions — sodium zirconium cyclosilicate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Chronic Kidney Disease patients not on dialysis: Chronic Kidney Disease patients not on dialysis
  Interventions: Drug: sodium zirconium cyclosilicate (SZC)
- Chronic Disease Patients on dialysis: Chronic Disease Patients on dialysis
  Interventions: Drug: sodium zirconium cyclosilicate (SZC)
- Heart Failure patients: Heart Failure patients receiving Renin angiotensin aldosterone inhibitors/Mineralocorticoid receptor antagonists (Raas i/Mras)
  Interventions: Drug: sodium zirconium cyclosilicate (SZC)

INTERVENTIONS:
Drug: sodium zirconium cyclosilicate (SZC) — sodium zirconium cyclosilicate (SZC), 5g or 10g of white to grey powder in a foil-lined packet. Starting dose of SZC is 10g, administered three times a day orally as a suspension in water. When normokalaemia has been achieved, starting dose of 5g once daily is recommended, with possible titration up to 10g once daily, or down to 5g once every other day, as needed, to maintain a normal potassium level. No more than 10g once daily should be used for maintenance therapy.

SUMMARY:
This is a multicenter, observational, prospective, national study which includes patients with chronic kidney disease (CKD) under dialysis or not, or with heart failure (HF), treated with sodium zirconium cyclosilicate (SZC) as per Summary of Product Characteristics (SmPC), aiming to collect information on patient characteristics, routine clinical practice and treatments administered for managing hyperkalaemia in a real-world setting in Greece. It will include approximately 12 public hospital and clinic based nephrology, or cardiology sites throughout the country. Sites and investigators will be selected so to represent the management of patients with CKD under dialysis or not, or with HF receiving Renin angiotensin aldosterone inhibitors/Mineralocorticoid receptor antagonists (RAASi/MRAs) therapy, and treated with sodium zirconium cyclosilicate (SZC) as per SmPC at a national level. The final selection of the participating sites will be based on a documented feasibility evaluation process that will assess physicians' qualifications, previous participation, and experience in similar clinical studies. Data will be obtained prospectively during the study visits as performed per standard clinical practice. Data regarding the patient's medical history will be collected retrospectively from patient medical charts records. Physicians will monitor eligible patients and will record their management according to their usual clinical practice. Only medical records available from the clinical practice and provided by the physicians will be used in this study as source documentation and the data will be entered into the electronic Case Report Form. Therefore, the collected data will reflect usual clinical practice. The study will enroll approximately 120 hyperkalaemia patients with serum potassium level >5.0 mmol/L, being treated with sodium zirconium cyclosilicate for hyperkalaemia at the time of enrolment as per SmPC, assigned in a 2:1:1 ratio to one of the following 3 groups: (1) CKD patients not on dialysis (60 patients), (2) CKD patients on dialysis (30 patients) and (3) HF patients receiving RAASi/MRAs therapy (30 patients), all consisting the study population. Patients will be followed for 6 months, with a 6-month recruitment period, for a total study duration of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form.
* Older than 18 years at the time of consent.
* Treated with sodium zirconium cyclosilicate (SZC) for hyperkalaemia at the time of enrolment, and having started receiving sodium zirconium cyclosilicate (SZC) at least 10 days before enrolment.
* Patients diagnosed with hyperkalaemia (Serum Potassium (S-K)+ >5.0 mmol/L), and with chronic kidney disease (CKD) not on dialysis (Group 1) or on dialysis (Group 2), or with heart failure (HF), receiving Renin angiotensin aldosterone inhibitors/Mineralocorticoid receptor antagonists (RAASi/MRAs) therapy (Group 3).

Exclusion Criteria:

* Patients who are pregnant, breast-feeding, or planning to become pregnant.
* Patients already participating in another clinical trial.
* Presence of a condition that, in the opinion of the investigator: i) would put the subject at undue risk, or ii) would potentially jeopardize the quality of the data to be generated, or iii) would, for some other reason, make the patient inappropriate for this study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 120 hyperkalaemia patients with serum potassium level >5.0 mmol/L, being treated with sodium zirconium cyclosilicate (SZC) for hyperkalaemia at the time of enrolment as per Summary of Product Characteristics (SmPC), assigned in a 2:1:1 ratio to one of the following 3 groups: (1) chronic kidney disease (CKD) patients not on dialysis (60 patients), (2) chronic kidney disease (CKD) patients on dialysis (30 patients) and (3) heart failure (HF) patients receiving Renin angiotensin aldosterone inhibitors/Mineralocorticoid receptor antagonists (RAASi/MRAs) therapy (30 patients)
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2024-02-09 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
To record the treatment patterns and characteristics of patients with hyperkalaemia receiving Sodium Zirconium Cyclosilicate (SZC) | Enrollment time point, 3 months after enrollment, 6 months after enrollment
  To describe the treatment patterns and patient characteristics of hyperkalaemia patients receiving Sodium Zirconium Cyclosilicate (SZC), by recording any pharmacological and other intervention administered, including dose and frequency of administration

CONTACTS AND LOCATIONS:
Locations (6):
- Greece (6):
  - Research Site, Alexandroupoli
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Larissa
  - Research Site, Pátrai
  - Research Site, Thessaloniki

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: CSR
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: D9480R00055_CSR Synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9480R00055&attachmentIdentifier=483d5244-08f6-4c46-8a5b-342b815b6942&fileName=D9480R00055_SHIELD_Clinical_Study_Report_Synopsis_final_22Dec2025_Redacted.pdf&versionIdentifier=